CLINICAL TRIAL: NCT06945614
Title: A Proof-of-Concept, Exploratory Clinical Study to Assess Safety and Efficacy of Xenon Gas Inhalation to Control Neuroinflammation in Healthy Human Subjects
Brief Title: Exploratory Clinical Study to Assess Safety and Efficacy of Xenon Gas Inhalation to Control Neuroinflammation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: General Biophysics LLC (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00082384; R42AG073059 (NIH); HLW-ALZ-Xen-001 (Other: FDA)
Record Dates: First submitted 2025-04-09; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer Study
Keywords: Xenon gas; inhalation; Alzheimer's disease; neurodegenerative; Healthy volunteer
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 10 minute inhalation (Experimental): Xenon gas inhalation administered for 10 minutes
  Interventions: Drug: Xenon gas inhalation
- 20 minute inhalation (Experimental): Xenon gas inhalation administered for 20 minutes
  Interventions: Drug: Xenon gas inhalation
- 30 minute inhalation (Experimental): Xenon gas inhalation administered for 30 minutes
  Interventions: Drug: Xenon gas inhalation
- 45 minute inhalation (Experimental): Xenon gas inhalation administered for 45 minutes
  Interventions: Drug: Xenon gas inhalation

INTERVENTIONS:
Drug: Xenon gas inhalation — Administration of xenon gas in the mixture with oxygen for the period of time via inhalation
  Other Names: Inhalation of xenon gas

SUMMARY:
The goal of this clinical study is to evaluate safety of Xenon gas inhalation in healthy volunteers. This first phase safety clinical study is part of evaluation of the xenon gas inhalation as a therapy for neurodegenerative diseases, such as Alzheimer's disease.

The investigators will administer xenon gas in low concentration to people via anesthetic machine, observe participants for sedation and any unexpected side effects, collect blood at each visit and measure the vital signs. There are four treatment groups in the study, which correspond with the duration of xenon gas treatment. Individual participation will last approximately 14 days over five visits: screening visit accompanied by the electrocardiogram, blood, and urine test; treatment visit for xenon gas inhalation treatment; and three follow up visits.

DETAILED DESCRIPTION:
The investigators plan to find out if xenon gas can help people with Alzheimer's disease, but it needs to be studied in healthy volunteers first. This study will show if xenon gas is safe to take without causing too many side effects. Xenon gas is not approved by the U.S. Food and Drug Administration (FDA). This means that the use of xenon gas is investigational and can only be used in research studies.

This single-center, open-label study will evaluate the safety and efficacy of xenon gas inhalation for 4 different durations of administration in healthy subjects. The study will be conducted at a single investigational site, with 4 dosing cohorts of 4 subjects each; xenon gas via inhalation for 10, 20, 30, and 45 minutes. Assignment into the study treatment groups occurs sequentially and participants will be informed which group they are in during the screening visit. This study will enroll healthy individuals who meet eligibility criteria. The maximum planned study duration for each subject is 15 days. This includes a screening period of up to 7 days during which eligibility is determined, and post-treatment observation on Days 1, 3 and 7 for follow-up safety monitoring.

Subjects will be screened and enrolled at the Center for Alzheimer Research and Treatment (CART). Initial treatment visits will occur in the Center for Clinical Investigation (CCI) with follow-up visits occurring in CART. Both centers are in the Building for Transformative Medicine, Brigham and Women's Hospital (BWH) at 60 Fenwood Road, Boston, MA 02115.

Participants will undergo screening procedures including hematology, clinical chemistry, vital signs, electrocardiogram (ECG), and a complete physical exam by the physician investigator or a mid-level practitioner. Each subject must have normal laboratory tests, or results must be in a clinically acceptable range in the opinion of the Investigator. Participants meeting eligibility criteria and completing screening activities will be assigned to a dosing group, based on the order of their enrollment after screening.

The dosing visit will occur the following week on a Monday or Tuesday. Participant's vital signs will be measured before study treatment administration, and on an ongoing basis throughout study treatment until discharged. Participant will also receive a dose of Zofran® prior to the administration of xenon gas to prevent any of the negative side effects that may occur. Xenon gas will be administered through machine providing gas inhalation (breathing in) under the supervision of a study anesthesiologist. An anesthesia face mask will be used to deliver the inhalation gas. The flow of xenon gas and oxygen will be controlled manually by the study anesthesiologist during the study treatment. The gas concentrations will be controlled and monitored by the study anesthesiologist. The monitors for blood pressure, pulse oximetry (measures blood oxygen), and electrocardiography (measures heart activity) will be attached to participant during the inhalation study treatment procedure. Participants will receive xenon gas inhalation for 10, 20, 30, or 45 minutes. After xenon gas inhalation, pure oxygen will be supplied for five minutes. The total procedure will take approximately 20 minutes longer than the specified administration period. Following dosing, participants will be monitored for at least 2 hours before being discharged. Additional blood sample and vitals will be obtained during monitoring.

Participants will make 3 additional visits; 1 day, 3 days, and 7 days following xenon gas administration. At each follow up visit, participants will undergo procedures including hematology, clinical chemistry, vital signs, ECG, and a complete physical exam by the physician investigator or a mid-level practitioner. Each subject must have normal laboratory tests, or results must be in a clinically acceptable range in the opinion of the Investigator. Blood samples for immunologic analysis will be obtained at every visit. Visit 5, or 7 days following xenon gas administration will be the final visit. After participants complete the study, they will be referred back to their own doctors for ongoing medical care.

ELIGIBILITY:
Inclusion Criteria:

Study subjects must meet the following eligibility criteria to participate in the study.

1. Male or female, aged 55-75 years.
2. Good general health with no disease likely to interfere with the study assessments.
3. Baseline vital signs within the following ranges:

   1. resting heart rate 60 to 90 BPM with Normal Sinus Rhythm
   2. respiratory rate less than 14
   3. resting diastolic blood pressure greater than 60 mm Hg and less than 90 mm Hg and resting systolic blood pressure less than 140 mm Hg and more than 110 mm Hg
   4. Peripheral blood oxygen saturation >95%
4. Immunizations fully up to date at Screening, according to the assessment of their primary care physician.
5. Negative urine pregnancy test within 7 days prior to the first dose of investigational product for women of childbearing potential, defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses any time in the preceding 24 consecutive months). Sexually active women of childbearing potential and male subjects must agree to use two effective contraceptive methods to avoid pregnancy (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for 90 days after the completion of study treatment. Contraceptive methods will be documented with other concomitant medications.
6. Willingness to comply with all study requirements.
7. Adequate cognitive function to understand and sign the IRB-approved ICF before any protocol-specific screening procedures are performed.

Exclusion Criteria:

Individuals who meet any of the following criteria at Screening will be excluded from the study:

1. Body mass index >30.
2. Any flu-like syndrome or other respiratory infections within 2 weeks prior to the Screening visit.
3. Active SARS-CoV-2 (COVID-19) disease.
4. A female who is pregnant, lactating, breastfeeding, or planning on becoming pregnant during study.

   1. Females of childbearing potential will undergo a pregnancy test at Screening and be excluded from the study if positive.
   2. A urine pregnancy test will also be performed on the morning of the dosing day.
5. History of a clinically significant acute or chronic disease that is not stable and medically managed in the judgment of the study physician.
6. History of bradycardia or other cardiovascular dysrhythmias or who are receiving beta blockers.
7. Cardiopulmonary disease, including pulmonary fibrosis, COPD, altered pulmonary function, lung injury, pulmonary hypertension, obstructive sleep apnea requiring CPAP.
8. Bowel obstruction, pneumocephalus, or other diseases with the potential for an air pocket and expansion following xenon administration.
9. Any medical condition or receiving any medications that predispose to delayed gastric emptying.
10. Known difficult airway, or potential for a difficult airway based on a thorough airway exam by an anesthesiologist.
11. Inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, asthma, thyroid disease, or type 1 diabetes.
12. Use of corticosteroids within the past month prior to the first treatment.
13. History of cancer in the past 5 years, with the exception of successfully treated basal cell carcinoma.
14. Any other clinically significant medical condition or illness as determined by medical history, clinical laboratory results, or other screening safety tests that, in the judgment of the Investigator, would interfere with participation in this study.
15. History of alcohol or substance abuse or dependence within the past 2 years.
16. Clinically significant abnormalities in screening laboratories.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Xenon Treatment-Related Adverse Events at Each Treatment Duration as Assessed by CTCAE v4.0 | From treatment to the end of follow up at 7 days
  To determine the safety of xenon gas inhalation for 10, 20, 30, and 45 minutes in healthy volunteers. Investigators anticipate to observe no sedation, no nausea, and no vomiting.
  Measured Parameters for Safety Assessments during Xenon Administration (Intraoperative - every five (5) minutes):
  * Heart rate
  * Blood pressure
  * Respiratory rate
  * Body temperature
  * Peripheral blood oxygenation
  * Changes in capnometry
  * Electrocardiographic parameters and printed rhythm strip
  * Adverse events Depth of sedation will be assessed and recorded every five (5) minutes during Xenon Gas administration and upon completion of procedure and recovery, utilizing the Modified Observer's Assessment of Alertness/Sedation Scale (MOAA/S) by the anesthesiologist. Adverse events of special interest for this inhaled anesthetic: vomiting, hemodynamic changes requiring drug intervention, and sedation unresponsive to verbal commands. AEs will be assessed during repeated visits on day 1, day 3, and day 7.

SECONDARY OUTCOMES:
Number of Participants With Treatment Related Change in Blood Biomarkers From the Baseline. | From treatment to the end of follow up in 7 days
  Depending on the duration of the xenon inhalation treatment and time after the treatment (immediately, 1 day, 3 days, and 7 days) the blood biomarkers will be measured. We anticipate to see the effect of xenon inhalation on immune cells as well as cytokines and hormones panels for the plasma samples. Specifically, the change from the baseline in the number and phenotypes of blood monocytes, Natural Killer Cells (NK), B cells, CD4, CD8 T cells and neutrophils will be measured. In addition the change from the baseline in cytokines and hormone levels in the plasma samples will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Ilin, PhD, Principal Investigator — General Biophysics; Howard L Weiner, MD, Principal Investigator — Brigham and Women"s Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandao W, Jain N, Yin Z, Kleemann KL, Carpenter M, Bao X, Serrano JR, Tycksen E, Durao A, Barry JL, Baufeld C, Guneykaya D, Zhang X, Litvinchuk A, Jiang H, Rosenzweig N, Pitts KM, Aronchik M, Yahya T, Cao T, Takahashi MK, Krishnan R, Davtyan H, Ulrich JD, Blurton-Jones M, Ilin I, Weiner HL, Holtzman DM, Butovsky O. Inhaled xenon modulates microglia and ameliorates disease in mouse models of amyloidosis and tauopathy. Sci Transl Med. 2025 Jan 15;17(781):eadk3690. doi: 10.1126/scitranslmed.adk3690. Epub 2025 Jan 15. PMID 39813317